CLINICAL TRIAL: NCT00348829
Title: Mitral Valve Reconstruction in Patients With Chronic Heart Failure and Secondary Mitral Insufficiency: Identification of Predictors for a Successful Therapy
Brief Title: Mitral Valve Reconstruction in Chronic Heart Failure (CHF): Identification of Predictors for a Successful Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: not enough patients to e recruited, problems with the conductance catheter
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Sven Möbius-Winkler, PD Dr. med., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: SMW 01
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2009-05

CONDITIONS: Chronic Heart Failure; Mitral Insufficiency
Keywords: CHF; mitral insufficiency; conductance catheter; mitral valve repair
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Surgical mitral valve reconstruction
  Interventions: Procedure: mitral valve repair
- 2 (No Intervention): conservative treatment

INTERVENTIONS:
Procedure: mitral valve repair — surgical mitral valve repair
  Arms: 1

SUMMARY:
The aim of the study is to evaluate hemodynamic and echocardiographic parameters in patients with secondary mitral insufficiency and CHF.

1. Identification of hemodynamic parameters as predictor for a successful mitral valve reconstruction in CHF patients.
2. Collection of clinical factors for the assessment of the postoperative course after mitral valve reconstruction in CHF patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Dilatative Cardiomyopathy with LVEF < 35%
3. NYHA III oder IV under maximal medical treatment
4. Angiographic and hemodynamic MI > II° (LAP- mean pressure > 15-20 mmHg; LA v-wave-oder PCWP v-wave > 35 mmHg under exercise)
5. Echocardiographic MI > II°
6. At least 1 hospitalization for heart failure before OP

Exclusion Criteria:

1. Secondary Cardiomyopathy by vitium cordis
2. Planned secondary procedure like CABG, aortic valve surgery, surgery of the tricuspid valve etc
3. Inclusion in another trial
4. Euro-Score > 30%
5. Former valve operation or CABG

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Identification of hemodynamic parameters as predictor for a successful mitral valve reconstruction in patients with congestive heart failure | 3 months

SECONDARY OUTCOMES:
Identification of clinical factors for the postoperative outcome | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schuler, Prof., Study Chair — Chair of the Dep. of Cardiology; Sven Möbius-Winkler, MD, Principal Investigator — Consultant of the dep. of Cardiology
Locations (1):
- Heart Center Leipzig GmbH, University Leipzig, Leipzig, Germany